CLINICAL TRIAL: NCT05029843
Title: Single Large-scale mtDNA Deletion Syndrome Natural History Study
Brief Title: SLSMDS Natural History Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Champ Foundation (Other)
Collaborators: Children's Hospital of Philadelphia (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: CFR-02
Record Dates: First submitted 2021-08-11; First posted 2021-09-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Pearson Syndrome; Single Large Scale Mitochondrial DNA Deletion Syndromes (SLSMDS)
MeSH Terms: conditions — VLCAD deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Single Large-Scale mtDNA Deletion Sydrome: Natural History Study (PS-NHS) aims to collect data on standardized clinical outcomes, store data on the Champ Foundation Registry (CFR) and make this data available to researchers, clinicians, and industry partners who are studying SLSMDS to answer questions regarding the disease, including its causes, potential treatments, and other topics. A secondary aim is to analyze the data to understand research questions relating to the natural history of SLSMDS.

DETAILED DESCRIPTION:
This study is a prospective, observational, and longitudinal study intended to track the course of Pearson syndrome and single large scale mitochondrial DNA deletion syndromes (SLSMDS) to identify demographic, genetic, environmental, and other variables that correlate with the diseases development and outcomes. If available, retrospective clinical data may be accessed and used in analyses as well.

The PS-NHS will be conducted at two Center of Excellence sites: the Cleveland Clinic and Children's Hospital of Philadelphia (CHOP).

All PS-NHS data will be entered and stored on the CFR. The CFR exists entirely online.

ELIGIBILITY:
Inclusion Criteria:

* Have an active account on the Champ Foundation Registry (CFR) or be willing to create an account on the CFR.
* Must have a genetic diagnosis of a single large-scale mitochondrial DNA deletion and must upload their genetic report to the CFR.
* Have a clinical diagnosis or history of Pearson syndrome OR have symptom onset prior to five years of age and a genetic diagnosis of a single large-scale mitochondrial DNA deletion OR in the opinion of the principal investigator the participant is suitable for participating in this study based on clinical presentation.

Participants may be of any age or gender, and originate from any country.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with confirmed Pearson Syndrome who satisfy the inclusion/exclusion criteria will be offered enrollment into this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-10-16 (Estimated); Study Completion 2024-10-16 (Estimated)

PRIMARY OUTCOMES:
Columbia Neurological Scale | 2 years
  The Columbia Neurological Scale is a neurological assessment that includes a general medical exam and a general neurological exam. It will take approximately 30 minutes to complete, and that includes evaluation of nerves, muscles and movement. Columbia Neurological Scale ranges from 0 (abnormal exam) to 76 (normal exam).
PEDI-CAT assessment | 2 years
  The PEDI-CAT is a computerized test that will ask participants about daily life tasks. This assessment will be given to patients 0 to 20 years old and will take approximately 15 minutes to complete.
International Pediatric Mitochondrial Disease Scale | 2 years
  The International Pediatric Mitochondrial Disease Scale is designed to monitor general disease progression associated with mitochondrial disease in children 0 to 18 years old. It includes a physical examination and evaluation of symptoms and functioning. The International Pediatric Mitochondrial Disease Scale will include a clinician-administered assessment that involves asking participants questions and evaluating participants' movements and responses, as well as a patient survey. The score is expressed as the percentage of items which were feasible to perform. Asterixes (*) can be scored as well, the total score will change accordingly. E.g. if the parents are not able to indicate the presence of headache, the maximum score of the first domain changes from 103 to 73. If the child is not cooperative during the execution of domain 2 and 3, these items are omitted from the total score.
Scale for Assessment and Rating of Ataxia | 2 years
  the SARA is a physical exam that evaluates symptoms of incoordination. A physician will complete this with exam and it will take approximately 20 minutes to complete.
Balance test | 2 years
  Standing balance test. May assessed with an accelerometer. Measured as time in seconds.
Coordination test | 2 years
  9-hold peg test. Measured as time in seconds.
2 or 6 minute walk test | 2 years
  2-minute walk test (2MWT) ages 3-6 yrs. or 6MWT (ages 6+). Measured as distance in meters.
Strength test | 2 years
  Hand grip with Dynamometer. Measured as average value of lbs of grip strength.
Hearing testing | 2 years
  Assessing hearing frequency in both ears.
EKG rhythm | 2 years
EKG PR interval | 2 years
EKG QRS interval | 2 years
Echo | 2 years
  Assessing valve abnormalities
BNP | 2 years
  Measured as pg/ml
Lipid panel | 2 years
  Total cholesterol, HDL-C, LDL-C, triglycerides. Measured as mg/dL.
Cortisol | 2 years
  Measured mcg/dL
PTH | 2 years
  Measured as pg/mL
Calcium | 2 years
  Measured as pg/mL
Vitamin D | 2 years
  Measured ng/mL
Growth hormone | 2 years
  Measured ng/mL
IGF1 | 2 years
  Measured ng/mL
TSH | 2 years
  Measured uIUg/mL
FT4 and T3 | 2 years
  Measured ng/dL
HbA1c | 2 years
  Measured as a percentage
C-peptide | 2 years
  Measured ng/mL
Fasting Plasma Glucose (FPG) | 2 years
  Measured mg/dL
Fructosamine | 2 years
  Measured mcmol/L
Amylase | 2 years
  Measured U/L
Comprehensive Metabolic Panel | 2 years
  Electrolytes, transaminases, TP/Albumin, bilirubin, alk phos, creatinine, BUN, GFR. Measured mmol/L.
Lipase | 2 years
  Measured U/L
PT/PTT | 2 years
  Measured in seconds
Stool elastase | 2 years
  ug Elastase/g stool
Height | 2 years
  Assessed in cm
Weight | 2 years
  Assessed in kg
Orbitofrontal cortex (OFC) | 2 years
  Assessed in cm
Complete blood count with differential | 2 years
Ferritin | 2 years
  Measured in ng/mL
Iron | 2 years
  Measured ug/dL
Reticulocytes | 2 years
  Count (x10^9/uL)
Reticulocytes | 2 years
  Percentage
Number of transfusions | 2 years
  Frequency count of number of red blood transfusions and platelet transfusions
Acylcarnitines (plasma) | 2 years
  Measured as mcmol/L
Amino acids (plasma and urine) | 2 years
  Interpretation recorded.
Organic acids (urine) | 2 years
  Interpretation recorded.
Lactate | 2 years
  measured mmol/L
Glutathione | 2 years
  Measured uM
GDF15 | 2 years
  pg/mL
Visual exam | 2 years
  Assessing palpebral fissure in mm; distance in mm; eye movement in mm
ERG/OCT | 2 years
  Assessed as normal or abnormal
Ptosis/ophthalmoplegia | 2 years
  Assessed in mm
Cystatin C | 2 years
  Measured mg/dL
Magnesium | 2 years
  Measured mg/dL
Phosphate | 2 years
  Measured mg/dL
Urine Electrolytes | 2 years
  Measured mg/dL
Urine protein | 2 years
  Measured mg/dL
Urine amino acids | 2 years
Facial dysmorphology assessment | 2 years
  Assessed with facial photography. Assessing ptosis and/or prominent cheeks/jowls.

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Parikh, MD, Principal Investigator — The Cleveland Clinic; Marni Falk, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
The data obtained during the study may be available on reasonable request.